CLINICAL TRIAL: NCT05045157
Title: Effectiveness of Percutaneous A1 Pulley Release Under Ultrasound Guidance Associated With Infiltration, Versus Infiltration Alone, in Patients With Trigger Finders Who Have Failed a First Infiltration: a Randomized Controlled Trial
Brief Title: Effectiveness of Percutaneous Pulley Release With Infiltration, Versus Infiltration Alone in Trigger Finders
Acronym: SECOIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHD21_0024
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutaneous A1 pulley release with corticosteroid injection (Experimental)
  Interventions: Procedure: Percutaneous A1 Pulley Release Under Ultrasound Guidance; Drug: Corticosteroid injection
- corticosteroid injection alone (Active Comparator)
  Interventions: Drug: Corticosteroid injection

INTERVENTIONS:
Procedure: Percutaneous A1 Pulley Release Under Ultrasound Guidance — the A1 pulley is cut off with Ultrasound guidance by a percutaneous insertion of the small needle under local anaesthesia.
  Arms: percutaneous A1 pulley release with corticosteroid injection
Drug: Corticosteroid injection — corticosteroid injection is performed

SUMMARY:
Trigger finger is a mechanical problem characterized by pain and catching of digit in flexion.

Histological changes of A1 pulley and synovial proliferation have been identified as factors that prompt trigger finger The first-line treatment of trigger finger is conservative with splinting and corticosteroid injection.

If the first infiltration fails, either a second infiltration or surgical sectioning of the pulley is proposed.

Surgery can be performed by several techniques (open section, percutaneous section with palpatory guidance, or under ultrasound guidance).

Percutaneous A1 pulley release under ultrasound guidance consists of cutting the A1 pulley by a percutaneous insertion with small needle under local anaesthesia.

The hypothesis of the study is that percutaneous A1 pulley release under ultrasound guidance followed by a corticosteroid injection would be more effective than a second corticosteroid injection alone on complete resolution of the trigger finger symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old,
* Presence of a trigger finger (thumb or long fingers) to be treated
* Quinnell score >1
* Episode of trigger characterized on questioning or clinical examination
* Failure of a first corticosteroid infiltration > 3 months before inclusion
* First infiltration within 15 months of inclusion
* Thickening A1 pulley on ultrasound ≥ 0.5 mm
* Patient who has the capacity to understand the protocol and has given consent to participate in the research,
* Patient with social security coverage

Exclusion Criteria:

* Presence of several symptomatic fingers requiring treatment by ultrasound-guided section of the pulley
* Patient who are pregnant, breastfeeding, or who have the potential to become pregnant without effective contraception at the time of inclusion
* Known allergy to corticoid (Hydrocortancyl®) including its excipients ((benzyl alcohol, sodium carmellose, sodium chloride, polysorbate 80)
* Known allergies to lidocaine
* Ongoing anticoagulant treatments (AVK, New Oral Anti-Coagulants)
* Local or general infection, or suspicion of infection
* Live vaccines
* Evolving viruses (hepatitis, herpes, varicella, shingles)
* Severe or uncontrolled hypertension
* Unbalanced diabetes
* Underlying progressive cardiovascular disease
* Hemodialysis patients
* Prosthesis on the finger to be treated
* Echographic tendon fissure
* Inflammatory disease (rheumatoid arthritis, spondyloarthritis, connective tissue diseases, etc.) with tenosynovitis.
* History of surgery on the fingers
* Dupuytren's disease
* Patient participating in another interventional clinical research protocol involving a drug or medical device
* Patient under guardianship, curators or legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of pulley section with ultrasound guidance combined with corticosteroid infiltration versus corticosteroid alone on complete resolution of trigger finger's symptoms | 1 year postoperatively
  Trigger finger's symptoms defined by a clinical Quinnell score ≤1 without the use of an alternative therapy

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Cormier, Dr, Principal Investigator — CHD Vendée
Locations (4):
- France (4):
  - Hopital Henri Mondor, Créteil
  - CHD Vendée, La Roche-sur-Yon
  - CHU Nantes, Nantes
  - Hopital Lariboisière, Paris

IPD SHARING:
Plan to Share IPD: No